CLINICAL TRIAL: NCT02592616
Title: Interval-training and Appetite Regulation in Patients With Type 2 Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Anders Rasmussen Rinnov, MD, PhD, Rigshospitalet, Denmark
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: H-15008542
Record Dates: First submitted 2015-10-28; First posted 2015-10-30 (Estimated); Last update posted 2016-06-22 (Estimated); Status verified 2016-06

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Exercise; Appetite; Energy intake
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- CON (Experimental): Control (CON).
  Interventions: Behavioral: CON
- CW (Experimental): Continuous Walking (CW).
  Interventions: Behavioral: CW
- IW (Experimental): Interval Walking (IW).
  Interventions: Behavioral: IW

INTERVENTIONS:
Behavioral: CON — No exercise intervention.
  Arms: CON
Behavioral: CW — One hour of continuous walking on a treadmill.
  Arms: CW
Behavioral: IW — One hour of interval (repeated cycles of 3 minutes of fast and 3 minutes of slow) walking on treadmill.
  Arms: IW

SUMMARY:
Four months of interval walking (IW) training results in substantial weight loss in opposition to energy-expenditure matched continuous walking (CW) training. The reason for this is unclear.

This study will assess if IW leads to greater exercise-induced suppression of appetite and ad libitum food intake compared to CW and no exercise.

Subjects with type 2 diabetes will be included in a crossover, counter-balanced, controlled study, where each subject will undergo three trials. Trials will be identical except the following interventions:

1. One hour of rest (CON)
2. One hour of interval walking (repeated cycles of 3 min of fast and 3 min of slow walking; IW)
3. One hour of continuous walking (CW) matched to IW with regards to energy-expenditure.

After the interventions subjects will undergo a liquid mixed meal tolerance test (450 kCal), with regular measurements of appetite-related hormones (insulin, ghrelin, Leptin, Cholecystokinin, PYY). Three hours into the mixed meal tolerance test, a standardised ad-libitum meal test will be served and intake will recorded. Free-living energy intake via food records will be assessed during the following 32 hours.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes Mellitus
* BMI > 25

Exclusion Criteria:

* Pregnancy
* Smoking
* Contraindication to increased levels of physical activity
* Eating disorder
* Insulin dependence

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2015-10; Primary Completion 2016-06 (Actual); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Ad-libitum meal energy intake | Initiated 3 hours after the intervention
  Subjects will receive a standardized ad-libitum meal and energy intake will be assessed

SECONDARY OUTCOMES:
Free-living energy intake | For 32 hours following the ad-libitum meal.
  Subjects will complete diet records for 32 hours following the ad-libitum meal and energy intake will be assessed.
Appetite-related hormones | Regularly during the 3 hours following the intervention
  Appetite-related hormones (insulin, ghrelin, leptin, cholecyctokinin, PYY) will be analysed in blood samples collected regularly during the liquid mixed-meal tolerance test following the intervention
Satiety | Regular assessments for 36 hours following the intervention
  Satiety questionaires will be completed at regular intervals after the intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Physical Activity Research (CFAS), Copenhagen, Denmark